CLINICAL TRIAL: NCT02635308
Title: Enhanced Rehabilitation Targeting Strength and Movement Pattern Symmetry Following Hip Fracture
Brief Title: Enhancing Rehabilitation After Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Robin Marcus, Ph.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00062639
Record Dates: First submitted 2015-11-30; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Hip Fracture
Keywords: hip fracture; physical function; muscle function; symmetry
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): High-Intensity, Unilaterally-Biased Resistance training 3x/wk x 12wk "MOVE"
  Interventions: Behavioral: Unilaterally Biased Resistance Training / "MOVE"

INTERVENTIONS:
Behavioral: Unilaterally Biased Resistance Training / "MOVE" — High-intensity resistance training including: whole body movement patterns, unilaterally biased lower extremity strength training, task-oriented balance tasks
  Other Names: High-Intensity Task Oriented Strength Training / "HI-TOSS"

SUMMARY:
This study evaluates the feasibility of implementing a unilaterally biased high-intensity resistance training to facilitate restorative vs. compensatory recovery after "usual care" physical therapy among older adults who have recently incurred a hip fracture. Additionally, physical performance during a sit-to-stand task, muscle function (strength/power), physical function measures, muscle composition, and muscle quality (force/unit area), are assessed before and after targeted high-intensity resistance training.

DETAILED DESCRIPTION:
Hip fracture is a major public health concern in the United States. Fall-related injuries constitute the leading cause of deaths and disabilities among persons over age 65 years. Hip fracture is consistently identified as one of the most frequent, costly, and devastating non-lethal injuries from a fall. Rehabilitation after hip fracture remains largely unchanged over the last 30 years despite evidence that high-intensity rehabilitation can benefit physical function after hip fracture beyond the recovery typical with "usual care".

Asymmetries demonstrated in physical performance of various tasks, such as gait, balance, and a sit-to-stand transfer, and impaired surgical limb muscle function are evident for years after hip fracture, and may contribute to the high rate of falls and declining function typically encountered by older adults recovering from hip fracture. Implementing a high-intensity rehabilitation approach targeting asymmetries after hip fracture is likely to yield improved symmetry in both physical function and muscle function. This study will recruit older adults who have recently incurred a hip fracture and completed "usual care" physical therapy to determine whether a high-intensity rehabilitation strategy targeting asymmetries in movement strategies and muscle function of the surgical limb can be successfully implemented in this challenging population. In particular, recruitment, adherence to rehab protocol parameters, and retention will be addressed among those who initiate high-resistance training at approximately 8-12wk after hip fracture incidence.

In addition, the investigators will explore the potential of targeted unilaterally-biased resistance training to improve surgical limb function and performance after hip fracture. Specifically, physical performance, muscle function, and muscle quality/composition are recorded and compared pre-/post-training to determine whether improvements occur in conjunction with high-intensity rehabilitation training. Additionally, the investigators will measure improvements in muscle composition that occur as a result of this high-intensity resistance training.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 50 yrs
* Ability to sign informed consent
* Mental Status MoCA score greater than 22
* Independent community ambulatory prior to hip fracture
* Ability to ambulate greater than 50 feet with or without assistive device

Exclusion Criteria:

* Previous hip fracture
* Bilateral hip fracture
* Pathological fracture
* Expected life Expectancy less than one year
* Permanently institutionalized
* Fracture result of multi-trauma
* Cardiac abnormalities
* Neuromuscular impairments
* Unstable medical conditions
* Elevated systolic greater than 150 or diastolic blood pressure greater than 100
* Implanted electronic devices
* History of stroke with motor disability
* Alcohol or drug abuse
* Respiratory disease
* Conditions deemed exclusionary by PI or physician

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
muscle strength | 12 week
  Knee extension muscle strength was measured on an isokinetic dynamometer as a maximum voluntary isometric contraction in newtons (N) of force. The average of three trials was used.
muscle power | 12 week
  Leg extension muscle power was measured on a Nottingham power rig in watts (W). The average of three trials was used.

SECONDARY OUTCOMES:
sit-to-stand task performance | 12 week
  biomechanics (vGRF) measured during sit-to-stand task performance
usual gait speed | 12 week
  Gait speed was measured at usual speed over a 50 foot distance and reported in meters/second.
muscle mass | 12 week
  MRI analysis of quadriceps muscle mass reported as average cross-sectional area in cm2.
Modified Physical Performance Test | 12 week
  The modified physical performance test (mPPT) is a standardized nine-item test designed to assess multiple dimensions of physical function was used to assess overall physical function. Scores are reported on a scale from 0-36.
Berg Balance Scale | 12 week
  The Berg Balance Scale (BBS) is a 14-item objective scale that provides a reliable and valid measure of static balance, with scores less than 45 indicating significant fall risk among older adults. Scores range from 0-56.
Timed up and Go Test | 12 week
  The Timed up and go test is recorded as the time in seconds to stand, walk 3 meters, turn around and return to a chair. The average time of three trials is reported.
Stair Climb Test | 12 week
  The time taken to ascend 10 stairs is reported.
Stair Descent Test | 12 week
  The time taken to descend 10 stairs is reported.
Lower Extremity Measure | 12 week
  The Lower Extremity Measure (LEM) is a 29-item self-report questionnaire that is reliable, valid, and responsive to improvement, with scores of 75 indicating moderate frailty, and scores above 85 indicating normal mobility and physical function after hip fracture. Scores range from 0-100.
Activities Specific Balance Scale | 12 week
  Activities-Specific Balance Confidence (ABC) scale is a 16-item, validated, reliable, self-report scale used to determine balance confidence. Scores range from 0-100.
Six minute walk test | 12 week.
  The distance in meters (m) walked in six minutes is recorded.

OTHER OUTCOMES:
muscle quality | 12 week
  muscle quality (force/unit area) calculated by using force and mass variables

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Marcus, PhD, Principal Investigator — University of Utah

REFERENCES:
- [Background] Kneiss JA, Houck JR, Bukata SV, Puzas JE. Influence of upper extremity assistance on lower extremity force application symmetry in individuals post-hip fracture during the sit-to-stand task. J Orthop Sports Phys Ther. 2012 May;42(5):474-81. doi: 10.2519/jospt.2012.3562. Epub 2012 Apr 30. PMID 22565360
- [Background] Kneiss JA, Hilton TN, Tome J, Houck JR. Weight-bearing asymmetry in individuals post-hip fracture during the sit to stand task. Clin Biomech (Bristol). 2015 Jan;30(1):14-21. doi: 10.1016/j.clinbiomech.2014.11.012. Epub 2014 Nov 29. PMID 25497603
- [Background] Edgren J, Rantanen T, Heinonen A, Portegijs E, Alen M, Kiviranta I, Kallinen M, Sipila S. Effects of progressive resistance training on physical disability among older community-dwelling people with history of hip fracture. Aging Clin Exp Res. 2012 Apr;24(2):171-5. doi: 10.1007/BF03325162. PMID 22842835
- [Background] Portegijs E, Kallinen M, Rantanen T, Heinonen A, Sihvonen S, Alen M, Kiviranta I, Sipila S. Effects of resistance training on lower-extremity impairments in older people with hip fracture. Arch Phys Med Rehabil. 2008 Sep;89(9):1667-74. doi: 10.1016/j.apmr.2008.01.026. PMID 18760151
- [Background] Portegijs E, Sipila S, Rantanen T, Lamb SE. Leg extension power deficit and mobility limitation in women recovering from hip fracture. Am J Phys Med Rehabil. 2008 May;87(5):363-70. doi: 10.1097/PHM.0b013e318164a9e2. PMID 18303470
- [Background] Edgren J, Salpakoski A, Rantanen T, Heinonen A, Kallinen M, von Bonsdorff MB, Portegijs E, Sihvonen S, Sipila S. Balance confidence and functional balance are associated with physical disability after hip fracture. Gait Posture. 2013 Feb;37(2):201-5. doi: 10.1016/j.gaitpost.2012.07.001. Epub 2012 Aug 9. PMID 22884315
- [Background] Host HH, Sinacore DR, Bohnert KL, Steger-May K, Brown M, Binder EF. Training-induced strength and functional adaptations after hip fracture. Phys Ther. 2007 Mar;87(3):292-303. doi: 10.2522/ptj.20050396. Epub 2007 Feb 6. PMID 17284548
- [Background] Binder EF, Brown M, Sinacore DR, Steger-May K, Yarasheski KE, Schechtman KB. Effects of extended outpatient rehabilitation after hip fracture: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):837-46. doi: 10.1001/jama.292.7.837. PMID 15315998
- [Background] Houck J, Kneiss J, Bukata SV, Puzas JE. Analysis of vertical ground reaction force variables during a Sit to Stand task in participants recovering from a hip fracture. Clin Biomech (Bristol). 2011 Jun;26(5):470-6. doi: 10.1016/j.clinbiomech.2010.12.004. Epub 2010 Dec 31. PMID 21196069
- [Background] Miller RR, Eastlack M, Hicks GE, Alley DE, Shardell MD, Orwig DL, Goodpaster BH, Chomentowski PJ, Hawkes WG, Hochberg MC, Ferrucci L, Magaziner J. Asymmetry in CT Scan Measures of Thigh Muscle 2 Months After Hip Fracture: The Baltimore Hip Studies. J Gerontol A Biol Sci Med Sci. 2015 Jun;70(6):753-6. doi: 10.1093/gerona/glr188. PMID 25958401
- [Background] D'Adamo CR, Hawkes WG, Miller RR, Jones M, Hochberg M, Yu-Yahiro J, Hebel JR, Magaziner J. Short-term changes in body composition after surgical repair of hip fracture. Age Ageing. 2014 Mar;43(2):275-80. doi: 10.1093/ageing/aft198. Epub 2013 Dec 25. PMID 24370941
- [Background] Penrod JD, Boockvar KS, Litke A, Magaziner J, Hannan EL, Halm EA, Silberzweig SB, Sean Morrison R, Orosz GM, Koval KJ, Siu AL. Physical therapy and mobility 2 and 6 months after hip fracture. J Am Geriatr Soc. 2004 Jul;52(7):1114-20. doi: 10.1111/j.1532-5415.2004.52309.x. PMID 15209649
- [Background] Magaziner J, Hawkes W, Hebel JR, Zimmerman SI, Fox KM, Dolan M, Felsenthal G, Kenzora J. Recovery from hip fracture in eight areas of function. J Gerontol A Biol Sci Med Sci. 2000 Sep;55(9):M498-507. doi: 10.1093/gerona/55.9.m498. PMID 10995047
- [Background] Visser M, Harris TB, Fox KM, Hawkes W, Hebel JR, Yahiro JY, Michael R, Zimmerman SI, Magaziner J. Change in muscle mass and muscle strength after a hip fracture: relationship to mobility recovery. J Gerontol A Biol Sci Med Sci. 2000 Aug;55(8):M434-40. doi: 10.1093/gerona/55.8.m434. PMID 10952365
- [Background] Fox KM, Magaziner J, Hawkes WG, Yu-Yahiro J, Hebel JR, Zimmerman SI, Holder L, Michael R. Loss of bone density and lean body mass after hip fracture. Osteoporos Int. 2000;11(1):31-5. doi: 10.1007/s001980050003. PMID 10663356